CLINICAL TRIAL: NCT00460369
Title: Sulfadoxine-Pyrimethamine Versus Artemether-Lumefantrine Versus Amodiaquine-Artesunate Coformulation in Uncomplicated Plasmodium Falciparum Malaria : an Open Randomized Study
Brief Title: Treatment of Uncomplicated Malaria in Benin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Faucher, Institut de Recherche pour le Développement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Malariallada
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Uncomplicated Malaria
Keywords: uncomplicated malaria; children; treatment; effectiveness
MeSH Terms: interventions — fanasil, pyrimethamine drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): sulfadoxine-pyrimethamine
  Interventions: Drug: sulfadoxine-pyrimethamine
- 2 (Active Comparator): artemether-lumefantrine
  Interventions: Drug: artemether-lumefantrine
- 3 (Active Comparator): amodiaquine-artesunate coformulation
  Interventions: Drug: amodiaquine-artesunate coformulation

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine — tablets 1,25/25 mg
  1 tablet per 20 kg of body weight Single drug intake
  Other Names: Fansidar
  Arms: 1
Drug: artemether-lumefantrine — tablets 20/120 mg
  * 1 tablet twice daily for 3 days below 15 kg of bodyweight
  * 2 tablets twice daily for 3 days below 24 kg of bodyweight
  * 3 tablets twice daily for 3 days below 35 kg of bodyweight
  Other Names: coartem
  Arms: 2
Drug: amodiaquine-artesunate coformulation — one 25mg/67,5mg tablet, once daily for 3 days below 9 kg
  one 50/135mg tablet, once daily for 3 days below 18 kg
  Other Names: coarsucam
  Arms: 3

SUMMARY:
Malaria is a life-threatening disease especially in small children. A high degree of Plasmodium falciparum resistance to chloroquine has already spread to South-Benin where this study is taking place. In the past few years, the recommendation for a first-line treatment in this area has moved from chloroquine to sulfadoxine-pyrimethamine (SP). There is growing evidence that Plasmodium falciparum resistance to SP has come to South-Benin. The aim of the study is to compare the efficacy of SP to two compact artemisinin-based therapies (ACT): artemether-lumefantrine and the amodiaquine-artesunate coformulation. ACT will be unsupervised.

The primary endpoint is an effectiveness comparison (PCR corrected) at day 28. Secondary outcomes are effectiveness comparisons (PCR corrected) at day 14 and 42 and a study on the relationships between ACT PK data (day 3) and outcome.

Expected total enrollment: 225 patients

Study start: April 2007; expected completion: December 2007

ELIGIBILITY:
Inclusion Criteria:

* 6-119 months old
* fever or history of fever of less than 24 hours
* p falciparum parasitemia > 1000 trophozoïtes/µL
* informed consent signed

Exclusion Criteria:

* < 5 kg
* danger or severity signs of malaria
* known underlying chronic disease
* Hb < 5g/dL
* adequate malaria treatment taken within 3 days before visit

Ages: 6 Months to 119 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
efficacy | day 28

SECONDARY OUTCOMES:
effectiveness comparisons (PCR corrected) | day 14 and day 42
incidence of adverse events | day 42

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Faucher, MD PhD, Principal Investigator — Institut de recherche pour le développement UR010; Philippe Deloron, MD PhD, Study Director — Institut de Recherche pour le Développement UR010
Locations (1):
- Centre de santé, Allada, Benin

REFERENCES:
- [Derived] Faucher JF, Aubouy A, Adeothy A, Cottrell G, Doritchamou J, Gourmel B, Houze P, Kossou H, Amedome H, Massougbodji A, Cot M, Deloron P. Comparison of sulfadoxine-pyrimethamine, unsupervised artemether-lumefantrine, and unsupervised artesunate-amodiaquine fixed-dose formulation for uncomplicated plasmodium falciparum malaria in Benin: a randomized effectiveness noninferiority trial. J Infect Dis. 2009 Jul 1;200(1):57-65. doi: 10.1086/599378. PMID 19469703